CLINICAL TRIAL: NCT03462901
Title: Fixation of Displaced Midshaft Clavicular Fractures in Adults by Intramedullary Elastic Rod
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrhman Ebrahem Kenan, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17100365
Record Dates: First submitted 2017-12-08; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Clavicular Fracture
Keywords: Fixation of midshaft clavicular fracture by intramedullary

STUDY DESIGN:
Intervention Model Description: Fracture clavicle in adults
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Elastic rod fixation (Experimental): Percutaneous intramedullary fixation of displaced midshaft clavicular fractures
  Interventions: Procedure: Percutaneous intramedullary fixation of displaced midshaft clavicular fractures .

INTERVENTIONS:
Procedure: Percutaneous intramedullary fixation of displaced midshaft clavicular fractures . — A group of 15 patients admitted to Assiut university with midshaft clavicular fractures treated by operative fixation of the fracture by single elastic rod through medial approach under image intensifier
  Other Names: Intramedulary fixation of clavicular fractures

SUMMARY:
Clavicular fracture, constitutes 2.6% e 5% of all adult fractures, most are located in the midshaft clavicle with different degrees of displacement. Conservative methods are commonly used for midshaft clavicular fractures treatment, but with various unsatisfactory complications such as nonunion, malunion and shoulders asymmetry. The rate of malunion after conservative treatment for the midshaft clavicular fractures reached 15%, and 30% patients were unsatisfied. Recently, early midshaft clavicular fractures could greatly reduce the incidence rate of nonunion and malunion. Open reduction and plate-screw ﬁxation was considered as the gold standard with the advantages of ﬁrm ﬁxation and earlier postoperative mobilization, but also with disadvantages of larger incision and more organizations being exposed, presenting with many postoperative complications. Intramedullary ﬁxation treatment for mid-clavicular fractures has been favored due to its strengths including small incision, less periosteal striping, dispersion of stress and simple to operate However, early intra-medullary implants, such as Hagie pins and Kirschner wires, have been gradually replaced due to insufficient stability. In addition, various nails such as elastic stable intramedullar

DETAILED DESCRIPTION:
Fixation of displaced midshaft clavicular fractures with minimally invasive technic as it helps for early mobilization to the shoulder and more safe, more cosmetically in comparison to other options.

ELIGIBILITY:
Adults pt aged (16-55 ) how is active presented with mid shaft clavicular fracture, displacement with no comorbidity and excluding pt with polytrauma aged above 55y or below 16y ,pt with fracture lateral 3rd and pt with comorbidity

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Male or female who is adult, active
Enrollment: 15 (Estimated)
Dates: Start 2016-10-30 (Actual); Primary Completion 2018-10-20 (Estimated); Study Completion 2019-05-21 (Estimated)

PRIMARY OUTCOMES:
Union rate | Six months
  We will compares rat of union between fixation of clavicular fracture by intramedullary elastic rod and other methods of fixation

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Fahmy Adam, Professor, Study Chair — Head of orthopedic and traumatology department

IPD SHARING:
Plan to Share IPD: Yes
Select patients and do the surgery and follow up prognosis
Supporting Information: Study Protocol
Time Frame: After six months
Access Criteria: Early preserve of shoulder activity